CLINICAL TRIAL: NCT01746927
Title: Does the Position of the Esophageal Entrance Determine the Cricoid Force Necessary to Occlude the Esophageal Lumen?
Brief Title: Does the Position of the Esophageal Entrance Determine the Cricoid Force Necessary to Occlude the Esophageal Lumen
Acronym: CP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Procare Riaya Hospital (Other)
Responsible Party: Principal Investigator, Ahed ZEIDAN, CONSULTANT ANESTHESIELOGIST, Procare Riaya Hospital
Other Study IDs: PRH05
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Aspiration
Keywords: cricoid pressure, glidescope

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cricoid pressure
  Interventions: Other: Glidescope Cricoid pressure

INTERVENTIONS:
Other: Glidescope Cricoid pressure — The current study test by direct visual evidence the occlusion of esophageal entrance during application CP. The closure of the lumen was further demonstrated by the inability to introduce a GT into the esophagus during CP. using in radimized method : 0 N,10 N, 20N AND 30 N

SUMMARY:
This investigation was designed to assess if the the position of esophageal entrance would detrmine the cricoid force necessary to occlude the esophageal lumen? in anesthetized, paralyzed non obese patients using the Glidescope ® video laryngoscope (GVL).

DETAILED DESCRIPTION:
80 adult patients (40 women, 40 men) scheduled to undergo elective surgical procedures requiring general anesthesia and necessitating endotracheal intubation, were included in this study. Patients eligible for participation were aged 18-60 yrs., ASA physical status I or II and BMI < 30 kg/m2. Before anesthesia induction, CP was verified as follow: the cricoid cartilage was first identified and then held between the thumb and middle finger and the pressure was applied by the index finger with a force that could be tolerated by the patient. After loss of consciousness, four predetermined forces: 0 , 10 , 20 and 30 N were chosen in a randomized method. Therefore, after applying the predetermined force, a GT 20 F insertion trial was performed and two outcomes were considered: 1) Failure of GT insertion: effective CP. The next trials were not attempted. 2) Success of GT insertion: ineffective CP. The patient received a second attempt with increasing force to the next scale of force. If the attempt was effective (failure of GT insertion) , the relevant force is considered as the effective CP force. Same trial was repeated using 0, 10, 20 and 30 N respectively in in a randomized fashion for each patient. The cricoid force was standardized by reproducing 10, 20 and 30 N on a weighing scale prior to each application.

Four anesthesia providers (operators) participated in the study: The first operator performed CP in all patients with his back towards the video monitor; the second operator performed laryngoscopy using GVL and GT insertion trials and he was not aware about the nature of study ; the third operator assessed the effectiveness of the applied CP and determined the position of the esophageal entrance in relation to the glottis. The fourth operator, who was standing behind the second operator, signaled to the second operator to start attempt for each trial with the predetermined CP forces and to the first operator who applying CP to stop or continue accordingly.

In order to "blind" the second operator, a screen separated the laryngoscopist and the first operator applying CP, while the hand position for the CP was maintained, even when CP was not applied. Data collected before staring surgery.

ELIGIBILITY:
Inclusion Criteria:

•No-obese patients (BMI < 30)

* ASA 1&2
* G.A needs intubation

Exclusion Criteria:

* ASA 3 and 4
* Contre indication to cricoid pressure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: normal healthy non obese patients
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Cricoid Pressure for Prevention of Aspiration | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ahed Zeidan, MD, Study Chair — Procare Riaya Hospital
Locations (1):
- Procare Riaya Hospital, Khobar, Estern, Saudi Arabia